CLINICAL TRIAL: NCT03477396
Title: A Phase IIA Trial Assessing the Tolerability of Ribociclib in Combination With an Aromatase Inhibitor in Patients Aged 70 and Older With Hormone Receptor Positive Metastatic Breast Cancer
Brief Title: Ribociclib and Aromatase Inhibitor in Treating Older Participants With Hormone Receptor Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17471; NCI-2018-00370 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17471 (Other: City of Hope Medical Center)
Record Dates: First submitted 2018-03-13; First posted 2018-03-26 (Actual); Results first posted 2022-05-18 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Estrogen Receptor and/or Progesterone Receptor Positive; HER2/Neu Negative; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: interventions — Aromatase Inhibitors; Pharmacogenomic Variants; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ribociclib, aromatase inhibitor) (Experimental): Participants receive ribociclib orally PO QD on days 1-21 and aromatase inhibitor per treating investigator's discretion. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Aromatase Inhibitor; Other: Laboratory Biomarker Analysis; Other: Pharmacokinetic Study; Other: Questionnaire Administration; Drug: Ribociclib

INTERVENTIONS:
Drug: Aromatase Inhibitor — Aromatase inhibitor per treating investigator's discretion
  Other Names: Androstenedione Aromatase Inhibitor; Estrogen Synthase Inhibitor; Estrogen Synthetase Inhibitor
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacokinetic Study — Correlative studies
  Other Names: PHARMACOKINETIC; PK Study
Other: Questionnaire Administration — Ancillary studies
Drug: Ribociclib — Given PO
  Other Names: Kisqali; LEE-011; LEE011

SUMMARY:
This phase IIA trial studies the side effects of ribociclib and aromatase inhibitor and how well they work in treating participants with hormone receptor positive breast cancer that has spread to other places in the body. Ribociclib and aromatase inhibitors may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the safety and tolerability of the combination of ribociclib and an aromatase inhibitor in adults age 70 or older with hormone receptor positive metastatic breast cancer.

SECONDARY OBJECTIVES:

I. To describe the full toxicity profile including all grades. II. To estimate the rate of worst grades of myelosuppression (neutropenia, leukopenia, thrombocytopenia, and anemia), neutropenic fever, gastrointestinal (GI) side effects (nausea, diarrhea, decreased appetite, vomiting, stomatitis), fatigue, neuropathy, and thromboembolism.

III. To describe rates of dose reductions, dose holds, and hospitalizations. IV. To estimate objective response rate and clinical benefit rate as defined by modified Response Evaluation Criteria in Solid Tumors (RECIST) (1.1) criteria.

V. To estimate median progression-free and overall survival.

EXPLORATORY OBJECTIVES:

I. To estimate the rate of adherence to ribociclib. II. To explore factors other than chronologic age that can affect toxicity rates as identified using a cancer-specific geriatric assessment.

III. To describe the results of the Was It Worth It (WIWI) and the results of the Overall Treatment Utility (OTU) Questionnaires.

OUTLINE:

Participants receive ribociclib orally (PO) once daily (QD) on days 1-21 and aromatase inhibitor per treating investigator's discretion. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 30 days, then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed the informed consent (ICF) prior to any study procedures being performed and is able to comply with protocol requirements
* Must be able to swallow ribociclib
* Age: >= 70 years at time of enrollment >= 70 to < 74 years, >= 75 years

  * NOTE: A minimum of 20 participants must be >= 75 years. The remaining 20 participants may be >= 70 to < 74 years OR >= 75 years
* Subjects must be able to communicate with the investigator and comply with the requirements of the study procedures
* Patient has a histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer, HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+, and metastatic breast cancer
* First or second line endocrine therapy for metastatic disease. One prior line of chemotherapy for metastatic disease is allowed
* Absolute neutrophil count >= 1.5 x 10^9 /L, at screening
* Platelets >= 100 x 10^9 /L, at screening
* Hemoglobin >= 9.0 g/dL, at screening
* Patient must have the following laboratory values within normal limits or corrected to within normal limits with supplement before the first dose of study medication:

  * Sodium
  * Potassium
  * Magnesium
  * Total calcium (corrected for serum albumin)
  * Phosphorous
* Serum creatinine < 1.5 mg/dL or creatinine clearance >= 50 mL/min, at screening
* In the absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x upper limit of normal (ULN); if the patient has liver metastases, ALT and AST < 5 x ULN, at screening
* Total bilirubin < ULN; or total bilirubin =< 3.0 x ULN or direct bilirubin =< 1.5 x ULN in patients with well-documented Gilbert's syndrome, at screening
* Patient with available standard 12-lead electrocardiogram (ECG) with the following parameters at screening (defined as the mean of the triplicate ECGs):

  * Fridericia's corrected QT (QTcF) interval at screening < 450msec (using Fridericia's correction)
  * Resting heart rate 50-90 beats per minute (bpm)

Exclusion Criteria:

* Patient received prior treatment with any CDK4/6 inhibitor
* Patient has a known hypersensitivity to any of the excipients of ribociclib
* Patients with a prior malignancy diagnosed within 2 years AND with evidence of disease (except adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer)
* Patient with concurrent malignancy that is not clinically stable AND needs tumor-directed therapy
* Patients with central nervous system (CNS) involvement unless they meet ALL the following criteria:

  * Untreated brain metastases (e.g., lesions < 1cm) not needing immediate local therapy
  * Previously treated brain metastases not needing immediate local therapy

    * At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment
    * Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormalities, including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to screening
  * Documented cardiomyopathy
  * Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block).
  * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

    * Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia
    * Concomitant use of medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued (within 5 half-lives or 7 days prior to starting study drug) or replaced by safe alternative medication
    * Inability to determine the QT interval on screening (QTcF, using Fridericia's correction)
  * Systolic blood pressure (SBP) > 160 mmHg or < 90 mmHg at screening
* Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to starting study drug:

  * Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pummelos, star-fruit, and Seville oranges
  * That have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
  * Herbal preparations/medications, dietary supplements
  * Warfarin or other coumadin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), newer anticoagulation agents such as direct factor Xa inhibitors, or fondaparinux is allowed
* Patient is currently receiving or has received systemic corticosteroids =< 2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment

  * The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular)
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.)
* Participation in a prior investigational study within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer
* Patient has had major surgery and/or radiotherapy within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery)
* Patient with a Child-Pugh score B or C
* Patient has not recovered from the acute effects of prior systemic therapy (until the toxicity resolves to either baseline or at least grade 1) except for residual alopecia or peripheral neuropathy
* Patient has a history of non-compliance to medical regimen or inability to grant consent
* Sexually active males unless they use a condom during intercourse while taking the drug and for 21 days after stopping treatment and should not father a child in this period; a condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2023-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mina Sedrak, MD, Principal Investigator — City of Hope Medical Center
Locations (9):
- United States (9):
  - City of Hope Corona, Corona, California
  - City of Hope Medical Center, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope Mission Hills, Mission Hills, California
  - City of Hope Rancho Cucamonga, Rancho Cucamonga, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope West Covina, West Covina, California
  - Roswell Park Cancer Institute, Buffalo, New York
  - Wilmot Cancer Institute, Rochester, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ribociclib, Aromatase Inhibitor)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ribociclib, Aromatase Inhibitor)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2
Karnofsky Status [Count of Participants; unit: Participants]
  100 - Normal no complaints; no evidence of disease | 1
  90 - Able to carry on normal activity; minor signs or symptoms of disease | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 2 and Above Toxicities Attributed to Ribociclib
Description: Number of participants with grade 2 and above toxicities attributed (possible, probable or definite) to ribociclib
Time Frame: Up to 30 days of last study drug, about 3 years and 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ribociclib, Aromatase Inhibitor)
Number analyzed (Participants) | 2
Participants | 2

2. Secondary Outcome: Number of Participants With Dose Reductions
Time Frame: Up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ribociclib, Aromatase Inhibitor)
Number analyzed (Participants) | 2
Participants | 2

3. Secondary Outcome: Number of Participants With Dose Delays
Time Frame: Up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ribociclib, Aromatase Inhibitor)
Number analyzed (Participants) | 2
Participants | 2

4. Secondary Outcome: Number of Participants With Dose Discontinuations
Time Frame: Up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ribociclib, Aromatase Inhibitor)
Number analyzed (Participants) | 2
Participants | 2

5. Secondary Outcome: Objective Response Rate by Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Objective response rate (defined as complete response [CR] + partial response [PR]) as determined by RECIST criteria
  Complete Response (CR): Disappearance of all target lesions. Lymph node CR is when the lymph node has decreased to less than 10mm in the short axis.
  Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ribociclib, Aromatase Inhibitor)
Number analyzed (Participants) | 2
Participants | 1

6. Secondary Outcome: Clinical Benefit Rate as Determined by RECIST
Description: Clinical benefit rate (defined as CR+PR+ stable disease) as determined by RECIST
  Complete Response (CR): Disappearance of all target lesions. Lymph node CR is when the lymph node has decreased to less than 10mm in the short axis.
  Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Up to 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ribociclib, Aromatase Inhibitor)
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Time Frame: Up to 30 days post cycle, up to 3.5 years total
Description: All serious adverse events are reported regardless of attribution and grade. Count of participants experiencing other adverse events are reported (after removing serious adverse from the toxicity dataset).
Arm/Group | Treatment (Ribociclib, Aromatase Inhibitor)
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ribociclib, Aromatase Inhibitor) (N=2)
Anemia (Blood and lymphatic system disorders) | 1
left upper eyelid droop (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 2
Pain (General disorders) | 1
Edema limbs (General disorders) | 1
blood in stool (General disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Cholesterol high (Investigations) | 1
Creatinine increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT03477396/Prot_SAP_000.pdf